CLINICAL TRIAL: NCT04828837
Title: National Taipei University of Nursing and Heath Sciences
Brief Title: Bubble PEP Training Among Patient With Chronic Obstructive Pulmonary Disease in Pulmonary Function Effects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the SARS-CoV-2 pandemic in Taiwan in 2021/05, and then recruitment was stopped under the government epidemic prevention policy.
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, SZU-YI WANG, Principal Investigator, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYWANG
Record Dates: First submitted 2021-02-25; First posted 2021-04-02 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: Chronic Obstructive Pulmonary Disease With Exacerbation; Chronic Obstructive Pulmonary Disease Exacerbation; Chronic Pulmonary Disease
Keywords: COPD, Bubble PEP, pulmonary function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bubble positive expiratory pressure training (Experimental): The experimental group receives the Bubble PEP training.
  Interventions: Device: bubble PEP
- general care (No Intervention): The control group receives the division of chest ward routine care.

INTERVENTIONS:
Device: bubble PEP — Using the bubble positive expiratory pressure (Bubble PEP) for breathing training of inpatients with COPD. The training course for one day of three times. Every time needs about 20 mins. Huff and cough after the breathing training the end.
  Arms: Bubble positive expiratory pressure training

SUMMARY:
The morbidity rate of Chronic Obstructive Pulmonary Disease (COPD) is increasing year by year. It is predicted to be the third leading cause of death worldwide in 2030. People with COPD have a high risk of needing a ventilator due to the decline of lung function, the increase of secretions, the dysfunction of airway clearance, and the obstruction and loss of alveolar elasticity.

DETAILED DESCRIPTION:
This study aimed to explore the effectiveness of cough and sputum assessment and respiratory physiological indicators after training with the Bubble positive expiratory pressure (Bubble PEP) inpatients with COPD. This is a randomization control trial design survey using convenient sampling and will be to select 94 inpatients with COPD in the division of chest ward of two teaching hospital in New Taipei City. The subjects who meet the conditions for admission are explained, and they need to sign a consent form confirming that they understand the risks. More, they are randomly divided into the experimental group (experimental group n=47) and the control group (control group n=47). The experimental group receives the Bubble PEP training; the control group receives the division of chest ward routine care. The study employs a structured questionnaire including a basic demography, COPD domain, COPD assessment test (CAT), cough and sputum assessment test, and check the peak expiratory flow rate (PEFR) using it for data collection. The study needs to be approve by the Institutional Review Board. The two groups agreed to participate in the study, after completing the subject consent form before the intervention, they also received the pre-test as a benchmark for the intervention effect. After completing the 7-day and 30-day intervention, the post-test was performed immediately to understand the intervention immediate effect.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients diagnosed with COPD
2. Over 40 years old
3. Awareness and ability to read articles
4. Agree to participate in this research and sign the research consent form

Exclusion Criteria:

1. Use non-invasive positive pressure breathing apparatus
2. Have received positive pressure breathing therapy before or during hospitalization
3. People with mental illness
4. Coughing up blood, pneumothorax
5. Suffer from legally infectious respiratory diseases
6. Pregnant women
7. Reject the subject

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Szu Yi Wang, Principal Investigator — none, specify Unaffiliated
Locations (1):
- National Taipei University of Nursing and Heath Sciences, Taipei, Beitou District, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study data were collected from February 2021 to July 2021 at two teaching hospitals in northern Taiwan.
Pre-assignment Details: In the study, 30 patients were excluded from the study before assignment to groups4 patients declined to participate, 10 inpatients had used non-invasive PEP treatment before hospitalization, 4 patients has a mental illness, and 12 patients have notifiable respiratory infectious diseases.
Period: Overall Study
Arm/Group | Bubble Positive Expiratory Pressure Training | General Care
Started | 13 | 14
Completed | 8 | 4
Not Completed | 5 | 10
Not completed — Stay-at-home during a COVID-19 outbreak | 1 | 3
Not completed — Lost to Follow-up | 2 | 6
Not completed — Lack of Efficacy | 1 | 0
Not completed — Admitted due to pneumothorax. | 1 | 0
Not completed — Admitted due to HIVD for operation. | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 27 participants in the study, 13 and 14 were assigned to the intervention and control groups, respectively. Two groups completed the sociodemographic characteristics and baseline test(T0).
Groups:
- Bubble Positive Expiratory Pressure Training; General Care: GOLD: Global Initiative for Chronic Obstructive Lung Disease; a Baseline (T0) data conduct homogenous test; Fisher's exact: Gander, Age, Marital status, Occupation, Smoking history, chronic comorbidities, diabetes mellitus, pneumothorax, lung cancer, COPD Grade
- Total: Total of all reporting groups
Arm/Group | Bubble Positive Expiratory Pressure Training | General Care | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Customized [Count of Participants; unit: Participants]
  Age : < 70 | 6 | 4 | 10
  Age : >= 70 | 7 | 10 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 14 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 13 | 14 | 27
Marital status [Count of Participants; unit: Participants]
  divorced/Single | 5 | 4 | 9
  married | 8 | 10 | 18
Occupation [Count of Participants; unit: Participants] — Blue-collar workers are individuals who perform hard manual labor in sectors such as agriculture, manufacturing, construction, mining, or maintenance.
  White-collar workers are typically found in office settings, characterized by their professional attire, often including white-collared shirts.
  Participants
    blue-collar worker | 7 | 10 | 17
    white-collar worker | 6 | 4 | 10
Smoking history [Count of Participants; unit: Participants]
  smoking | 3 | 4 | 7
  non-smoking | 1 | 1 | 2
  quit-smoking | 9 | 9 | 18
Chronic comorbidities [Count of Participants; unit: Participants]
  Hypertension | 6 | 7 | 13
  Diabetes mellitus | 1 | 2 | 3
  Heart disease | 6 | 6 | 12
  Pneumothorax | 0 | 2 | 2
  Lung cancer | 1 | 0 | 1
COPD Grade [Count of Participants; unit: Participants]
  GOLD 2(FEV1 50-79) | 2 | 6 | 8
  GOLD 3(FEV1 30-49) | 11 | 8 | 19
Dry powder bronchodilator use (day) [Mean (Standard Deviation); unit: days] | 7.25 (4.31) | 3.30 (2.41) | 5.45 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: The Chinese Version of Chronic Obstructive Pulmonary Disease Assessment Test(CAT)
Description: In the CAT, a total of eight items were used to assess the degree of dyspnea of the patients. Each item had a score ranging from 0 to 5 points, with the lowest total score being 0 points and the highest total score being 40 points. The higher the score, the higher the degree of dyspnea.
Time Frame: The pre-tests within 48 hours of hospitalization, which served as the baseline of the intervention (T0). Assessed at 1(T1) and 4(T2) weeks, week 4 was reported.
Population: A total of 57 were randomly assigned and complete test, with 13 in the experimental group and 14 in the control group. At T1, the experimental group had 11 analyzed, experiencing a total loss of 2 participants. In comparison, the control group had 6 analyzed at T1, with a cumulative loss of 8 participants. Moving to T2, the experimental group had 8 analyzed, with a total loss of 3 participants. The control group had 4 analyzed at T2, with a cumulative loss of 2 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- General Care Group: A total of 14 participants were enrolled in the control group and completed the baseline CAT (T0). After 7 days, in the second round, 6 participants completed the CAT T1 assessment. Five participants refused to participate in the breathing training, one participant was hospitalized for treatment due to a herniated disc, and one participant was unable to complete the T1 assessment as they stayed at home during the COVID-19 outbreak. After a 30-day study period, in the third round (T2), 6 participants completed the assessment. Two participants did not complete the third assessment. Among the participants who did not complete the third assessment, one individual refused further breathing training, and one individual stayed at home during the COVID-19 outbreak.
- Intervention Group: A total of 13 participants were enrolled in the intervention group and completed the baseline CAT (T0). After 7 days, in the second round, 11 participants completed the CAT T1 assessment. Two participants were unable to complete the T2 assessment due to their inability to learn breathing techniques. After a 30-day study period, in the third round (T2), 8 participants completed the assessment. Among the participants who did not complete the third assessment, one individual refused to participate in the breathing training, one was hospitalized due to spontaneous pneumothorax, and one stayed at home during the COVID-19 outbreak.
Arm/Group | General Care Group | Intervention Group
Number analyzed (Participants) | 14 | 13
score on a scale
  T0 | 13 (6.33) | 19.77 (6.26)
  T1: number analyzed (Participants) | 11 | 6
  T1 | 11.17 (8.04) | 13.18 (10.59)
  T2: number analyzed (Participants) | 8 | 4
  T2 | 9.50 (9.26) | 9.63 (6.78)
Statistical Analysis 1: Comparison: General Care Group vs Intervention Group; Descriptive statistics, including count, percentage, mean, and standard deviation, were used to summarize the data; Test type: Superiority — The intervention effect was evaluated using the generalized estimating equation (GEE) statistical method. Two-tailed tests were conducted, and p-values less than .05 were considered statistically significant; p < 0.05, Wilcoxon (Mann-Whitney) — We used Mann-Whitney U test for independent samples, and Fisher's exact tests when more than 20% of cells have expected frequencies <5 or less than 10 observations to examine the homogeneity between groups based on demographic characteristics; Mean Difference (Final Values) = 0.39

2. Primary Outcome: The Cough With Sputum Symptoms Assessment Questionnaire(CSSAQ)
Description: CSSAQ is used to assess patients' cough and sputum symptoms. The questionnaire content is based on published literature. It consists of 25 questions, including issues related to cough, sputum, and psychological symptoms and impacts. The scoring uses a four-point Likert scale, with scores ranging from 0 to 4, where higher scores indicate more severe symptoms. The total scale score ranges from a minimum of 0 to a maximum of 100. The content validity index is 1, and the Cronbach's α is 0.97.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Bubble Positive Expiratory Pressure Training: A total of 13 participants were enrolled in the intervention group and completed the baseline C (T0). After 7 days, in the second round, 11 participants completed the CASSAQ T1 assessment. Two participants were unable to complete the T2 assessment due to their inability to learn breathing techniques. After a 30-day study period, in the third round (T2), 8 participants completed the assessment. Among the participants who did not complete the third assessment, one individual refused to participate in the breathing training, one was hospitalized due to spontaneous pneumothorax, and one stayed at home during the COVID-19 outbreak.
- General Care: A total of 14 participants were enrolled in the control group and completed the baseline CASSAQ (T0). After 7 days, in the second round, 6 participants completed the CASSAQ T1 assessment. Five participants refused to participate in the breathing training, one participant was hospitalized for treatment due to a herniated disc, and one participant was unable to complete the T1 assessment as they stayed at home during the COVID-19 outbreak. After a 30-day study period, in the third round (T2), 6 participants completed the assessment. Two participants did not complete the third assessment. Among the participants who did not complete the third assessment, one individual refused further breathing training, and one individual stayed at home during the COVID-19 outbreak.
Arm/Group | Bubble Positive Expiratory Pressure Training | General Care
Number analyzed (Participants) | 13 | 14
score on a scale
  T0 | 14.38 (10.46) | 27.00 (23.31)
  T1: number analyzed (Participants) | 11 | 6
  T1 | 23.64 (20.92) | 29.83 (28.34)
  T2: number analyzed (Participants) | 8 | 4
  T2 | 14.38 (10.46) | 27.00 (23.31)
Statistical Analysis 1: Comparison: Bubble Positive Expiratory Pressure Training vs General Care; Descriptive statistics, including count, percentage, mean, and standard deviation, were used to summarize the data; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.05, The generalized estimating equation (GEE — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Peak Expiratory Flow Rate(PEFR)
Description: The TruZone peak flow meter is used to monitor the patient's Forced Expiratory Volume in the first second (FEV1). For each data collection session, three maximum expiratory flow tests are conducted, and the best value is taken as the result for that session. The measurement unit is ml/sec.
Time Frame: The study lasted 30 days with a total of three measurements. The first measurement baseline was 48 hours after hospitalization, the second on day 7 of the study, and the third on day 30 of the study.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml/sec
Groups:
- Bubble Positive Expiratory Pressure Training: A total of 13 participants were enrolled in the intervention group and completed the baseline PEFR (T0). After 7 days, in the second round, 11 participants completed the PEFR T1 assessment. Two participants were unable to complete the T2 assessment due to their inability to learn breathing techniques. After a 30-day study period, in the third round (T2), 8 participants completed the assessment. Among the participants who did not complete the third assessment, one individual refused to participate in the breathing training, one was hospitalized due to spontaneous pneumothorax, and one stayed at home during the COVID-19 outbreak.
- General Care: A total of 14 participants were enrolled in the control group and completed the baseline PEFR (T0). After 7 days, in the second round, 6 participants completed the PEFRT1 assessment. Five participants refused to participate in the breathing training, one participant was hospitalized for treatment due to a herniated disc, and one participant was unable to complete the T1 assessment as they stayed at home during the COVID-19 outbreak. After a 30-day study period, in the third round (T2), 6 participants completed the assessment. Two participants did not complete the third assessment. Among the participants who did not complete the third assessment, one individual refused further breathing training, and one individual stayed at home during the COVID-19 outbreak.
Arm/Group | Bubble Positive Expiratory Pressure Training | General Care
Number analyzed (Participants) | 13 | 14
ml/sec
  T0 | 320.00 (94.57) | 232.50 (85.00)
  T1 | 250.45 (82.60) | 273.33 (89.14)
  T2 | 320.00 (94.57) | 232.50 (85.00)
Statistical Analysis 1: Comparison: Bubble Positive Expiratory Pressure Training vs General Care; Descriptive statistics, including count, percentage, mean, and standard deviation, were used to summarize the data; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.05, The generalized estimating equation (GEE — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Re-hospitalization Event
Description: The number of patients who were readmitted due to COPD acute exacerbation (COPDAE) within 14 days after discharge during the study.
Time Frame: Within 14 days after discharge.
Measure: Number; unit: Number
Groups:
- Bubble Positive Expiratory Pressure Training: During the study, no patients in the experimental group were readmitted due to COPD acute exacerbation within 14 days after discharge.
- General Care: During the study, no patients in the control group were readmitted due to COPD acute exacerbation within 14 days after discharge.
Arm/Group | Bubble Positive Expiratory Pressure Training | General Care
Number analyzed (Participants) | 8 | 6
Number
  rehospitalization event | 0 | 0
  non rehospitalization event | 8 | 6
Statistical Analysis 1: Comparison: Bubble Positive Expiratory Pressure Training vs General Care; Test type: Superiority; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 30 days
Description: The possible adverse reaction in this study is hyperventilation, and its symptoms are dizziness, headache, nausea, blurred vision, rapid heartbeat, skin heat, muscle cramps, etc.
Groups:
- Bubble Positive Expiratory Pressure Training: Denied any adverse event in the experimental group.
- General Care: Denied any adverse event in the control group.
Arm/Group | Bubble Positive Expiratory Pressure Training | General Care
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

LIMITATIONS AND CAVEATS:
This study was affected by the COVID-19 pandemic. Due to the high attrition rate, our ITT results may have led to over- or underestimation of the effectiveness of the intervention. Sample size should therefore be increased in future studies. In addition, we used self-administered questionnaires for all measures except the PEFR test to evaluate intervention effectiveness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT04828837/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT04828837/SAP_001.pdf